CLINICAL TRIAL: NCT02975479
Title: Intralymphatic Immunotherapy in Increasing Doses up to 10 000 SQ-U - a Human Randomized Clinical Trial. Substudy.
Brief Title: Intralymphatic Immunotherapy in Increasing Doses, Substudy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Skane University Hospital (Other); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Lars Olaf Cardell, Professor, Head of Division, M.D., Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-001259-63 substudy
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2020-10

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Hay fever; Pollen allergy; Allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — Allergens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intralymphatic placebo injections (Placebo Comparator): ALK Diluent, ATC-code V07AB. 3 injections with 4-7 weeks interval.
  Interventions: Drug: ALK Diluent
- Intralymphatic active injections (Active Comparator): ATC-code V01AA02. 3 injections with 4-7 weeks interval in an up-dosing protocol; 1000 SQ-U, 3000 SQ-U, 10000 SQ-U.
  ***IMPORTANT INFORMATION! The up-dosing protocol is changed due to an adverse event at the last injection. New regimen: 1000 SQ-U, 3000 SQ-U, 3000 SQ-U. ***
  Interventions: Drug: ALK Alutard SQ 5-grasses or ALK Alutard Birch

INTERVENTIONS:
Drug: ALK Diluent
  Other Names: 0,3% human albumin. ATC-code V07AB
  Arms: Intralymphatic placebo injections
Drug: ALK Alutard SQ 5-grasses or ALK Alutard Birch — Depot formulation of relevant allergen adsorbed to aluminium hydroxide in a suspension.
  Other Names: Allergen, grass pollen. ATC-code V01AA02 or V01AA05
  Arms: Intralymphatic active injections

SUMMARY:
The study evaluates the safety and effect of intralymphatic allergen specific immunotherapy in increasing doses. Patients with allergy to grass or birch will be treated with three intralymphatic injections in an up-dosing protocol; 1000 SQ-U, 3000 SQ-U and 10 000 SQ-U, or placebo.

***IMPORTANT INFORMATION!*** The up-dosing protocol is changed due to adverse events at 5000 SQ-U. One patient had general utricaria 15 minutes after injection (moderate reaction). One patient had a serious adverse event with anaphylactic reaction 6 minutes after intralymphatic injection. (1000 SQ-U and 3000 SQ-U have been given with no serious adverse events.) New regimen: 1000 SQ-U, 3000 SQ-U, 3000 SQ-U.

DETAILED DESCRIPTION:
40 patients with seasonal allergic rhinitis will be recruited. Study subjects are randomized to intralymphatic injections with placebo or ALK Alutard 5-grasses or birch. Injections are given with 4-5 (-7) weeks interval.

ELIGIBILITY:
Inclusion Criteria:

* Seasonal allergic symptoms for birch and/or grass verified by skin prick test,
* Accepted informed consent

Exclusion Criteria:

* Pregnancy or nursing
* Autoimmune or collagen disease (known)
* Cardiovascular disease
* Perennial pulmonary disease
* Hepatic disease
* Renal disease
* Cancer
* Any medication with a possible side-effect of interfering with the immune response
* Previous immuno- or chemotherapy
* Chronic diseases
* Other upper airway disease (non-allergic sinusitis, nasal polyps, chronic obstructive and restrictive lung disease)
* Disease or conditions rendering the treatment of anaphylactic reactions difficult (symptomatic coronary heart diseases, severe arterial hypertension and treatment with β-blockers)
* Major metabolic disease
* Known or suspected allergy to the study product
* Alcohol or drug abuse
* Mental incapability of coping with the study
* Withdrawal of informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-05; Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Mean combined daily symptoms-and-medications-score | Peak pollen season (approximately 6 months after completed treatment) and entire pollen season (5-7 months after treatment).
  Daily scoring of rhinoconjunctivitis symptoms (6 questions, 4-point scale) and medication use (oral or topical antihistamines, intranasal corticosteroids, oral corticosteroids).

SECONDARY OUTCOMES:
Mean total daily symptoms score | Peak pollen season (approximately 6 months after completed treatment) and entire pollen season (5-7 months after treatment).
  Daily scoring of rhinoconjunctivitis symptoms (6 questions, 4-point scale)
Mean total daily medications score | Peak pollen season (approximately 6 months after completed treatment) and entire pollen season (5-7 months after treatment).
  Daily scoring of medication use (oral or topical antihistamines, intranasal corticosteroids, oral corticosteroids).
Change in subjective allergic symptoms following nasal allergen provocation | Before treatment, an average of 4 weeks after completed treatment and 6-9 months after treatment.
  The study subjects will be intranasally challenged with allergen and symptom score questionnaires are filled out pre-provocation and 5, 10 and 30 min post-provocation.
Effects on quality of life | During peak pollen season which will be up to 6 months after completed treatment.
  Juniper Rhinitis quality of life questionnaire (RQLQ) questionnaires
Short term change of skin reactivity | Before treatment, an average of 4 weeks after completed treatment and 6-9 months after treatment.
  Skin prick test
S-IgE Grass or Birch | Before treatment, approximately 4 weeks after completed treatment and 6-9 months after treatment
S-IgG4 Grass or Birch | Before treatment, approximately 4 weeks after completed treatment and 6-9 months after treatment
Registration of adverse event | From the first injection to 30 days after the last injections has been given

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Olaf Cardell, Professor, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Allergic Unit at the Department of Oto-Rhino-Laryngology at Skåne University Hospital Lund, Lund
  - ENT-department, Karolinska University Hospital Huddinge (ENT-department B51), Stockholm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hellkvist L, Hjalmarsson E, Weinfeld D, Dahl A, Karlsson A, Westman M, Lundkvist K, Winqvist O, Georen SK, Westin U, Cardell LO. High-dose pollen intralymphatic immunotherapy: Two RDBPC trials question the benefit of dose increase. Allergy. 2022 Mar;77(3):883-896. doi: 10.1111/all.15042. Epub 2021 Aug 29. PMID 34379802